CLINICAL TRIAL: NCT06621173
Title: A Clinical Trial Assessing the Safety and Efficacy of Intravenous HNF4α SrRNA for the Treatment of Patients With Metastatic Colorectal Cancer
Brief Title: A Clinical Trial Evaluating the Safety and Efficacy of Intravenous HNF4α SrRNA in Treating Metastatic CRC Patients
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Wei-Fen Xie, Director, Department of Gastroenterology, Changzheng Hospital, Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZXH-CRC-2024-IIT
Record Dates: First submitted 2024-09-24; First posted 2024-10-01 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Colorectal Cancer (mCRC)
Keywords: colorectal cancer; Hepatocyte nuclear factor 4α
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: The subjects with metastatic colorectal cancer will be treated by HNF4α srRNA intravenously via a peripheral vein.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HNF4α srRNA treatment (Experimental): The subjects with metastatic colorectal cancer will be treated by HNF4α srRNA intravenously via a peripheral vein.
  According to Amendment 1, the HNF4α srRNA preparation CD-801 used in the original protocol will expire on December 31, 2024. For participants receiving treatment after this date, the preparation will be switched to CD-GA-102, with the treatment dose converted on a 1:1 basis.
  Interventions: Drug: HNF4α srRNA

INTERVENTIONS:
Drug: HNF4α srRNA — HNF4α srRNA will be administered intravenously for the treatment of metastatic colorectal cancer. The dosing regimen is planned for a second dose 14 ± 3 days post-initial treatment, followed by subsequent treatments every 28 ± 7 days, with adjustments made based on patient tolerance and therapeutic response.
  According to Amendment 1, after enrollment, the investigator will determine the HNF4α srRNA dose, whether to combine it with immunotherapy, and the dose and schedule of the combination, based on the patient's treatment history and the safety/efficacy data of HNF4α srRNA administered via peripheral vein for hepatocellular carcinoma, intrahepatic cholangiocarcinoma, or colorectal cancer. Participants initially on HNF4α srRNA monotherapy who are considered for combination with immunotherapy must complete at least two treatment cycles and the post - treatment safety assessment.

SUMMARY:
This trial is a single-arm, open-label, exploratory first-in-human clinical study designed to evaluate the safety and tolerability of HNF4α srRNA injection in patients with locally unresectable or metastatic colorectal cancer, and to preliminarily explore its effectiveness in treating metastatic colorectal cancer.

DETAILED DESCRIPTION:
This study will administer HNF4α srRNA via intravenous injection to treat locally unresectable or metastatic colorectal cancer. The second treatment will be conducted 14 ± 3 days after the initial treatment, with subsequent treatment cycles every 28 ± 7 days (the dosing interval will be adjusted based on the tolerability, safety, and therapeutic effect of the subjects). The dose-escalation trial will employ the i3+3 design method, with three dose groups, tentatively setting the injection dose of HNF4α srRNA at 25 μg, 50 μg, and 100 μg per administration, and each group is expected to include up to 3 subjects.

According to Amendment 1, after enrollment, the investigator will determine the HNF4α srRNA dose, whether to combine it with immunotherapy, and the dose and schedule of the combination, based on the patient's treatment history and the safety/efficacy data of HNF4α srRNA (CD-801/CD-GA-102) administered via peripheral vein for hepatocellular carcinoma (HCC), intrahepatic cholangiocarcinoma (ICC), or colorectal cancer (CRC). Participants initially on HNF4α srRNA monotherapy who are considered for combination with immunotherapy must complete at least two treatment cycles and the post - treatment safety assessment. Then, the investigator can decide whether to add immunotherapy after a comprehensive review of their treatment history.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, aged 18 years or older.
2. Patients with histologically confirmed colorectal cancer that has been determined to be unresectable or metastatic.
3. Colorectal cancer subjects who are unsuitable or unable to tolerate standard systemic therapy, or who have received standard systemic therapy but have disease progression based on RECIST (version 1.1) criteria, including chemotherapy based on fluorouracil, oxaliplatin, or irinotecan, and targeted therapies with anti-VEGF/EGFR monoclonal antibodies.
4. Patients with confirmed deficient mismatch repair (dMMR) or high microsatellite instability (MSI-H) in tumor tissue, who have been treated with immune checkpoint inhibitors (anti-PD-1 or anti-PD-L1 antibodies) and are assessed with disease progression.
5. According to the RECIST (version 1.1) criteria, there are measurable target lesions suitable for repeated measurements for assessment.
6. Life expectancy of 12 weeks or more.
7. Subjects must have an Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 to 2.
8. Males with fertility and females of childbearing potential are willing to use a highly effective method of contraception for the entire study period and for 6 months after study drug discontinuation. Females of childbearing age, including premenopausal females and within 2 years after menopause, must have a negative serum pregnancy test result within 7 days prior to the first dose of study treatment.
9. Subjects who had a voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol.

Exclusion Criteria:

* Patients with any of the following criteria were excluded from participation in this study

  1. Patients who have undergone standard adjuvant chemotherapy after tumor resection, and have experienced recurrence or metastasis within 6 months after discontinuing the medication, and have not received standard systemic therapy.
  2. Clinical or imaging indications suggest the current presence of intestinal obstruction, perforation, or bleeding; or those who, upon investigator assessment, are at a higher risk of perforation or bleeding.
  3. Inadequate liver function：serum bilirubin > 3 × the upper limit of normal (ULN), or aspartate aminotransferase (AST), alkaline phosphatase (ALP), or alanine aminotransferase (ALT) > 5 × ULN.
  4. Inadequate renal function defined as creatinine >1.5 × ULN or calculated creatinine clearance < 40 mL/min.
  5. Absolute neutrophil count (ANC) < 1.5×109/L, or Platelets < 50×109/L, or Hemoglobin < 9.0 g/dL.
  6. International normalized ratio (INR) > 2.0.
  7. Patients with confirmed tumor brain metastases.
  8. Poorly controlled hypertension, diabetes or other serious heart or lung diseases, or with serious dysfunction.
  9. Patients who have received local or systemic anti-tumor treatments such as immunotherapy, targeted therapy, and chemotherapy within 4 weeks, or radiation therapy within 3 weeks, except for treatment regimens assessed as disease progression according to RECIST v1.1.
  10. All toxicities related to prior locoregional or systemic anti-tumor treatments are still grade 2 or more (except for hair loss and other events that have been judged tolerable by researchers).
  11. Uncontrolled active infection (eg, lung infections, or abdominal infections).
  12. History of malignancy other than CRC within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year overall survival rate > 90%), such as adequately treated early gastric carcinoma, carcinoma in situ of the cervix, non-melanoma skin carcinoma, or localized prostate cancer.
  13. Having an active autoimmune disease that requires systemic treatment within the past 2 years.
  14. Any condition requiring systemic treatment with corticosteroids (prednisone or equivalent >10mg/day) or other immunosuppressive drugs within 14 days prior to the first administration of the investigational drug.
  15. Patients with a history of organ transplantation.
  16. Hepatitis B virus DNA greater than 500 IU/ml, or hepatitis C virus RNA greater than 100 IU/ml.
  17. Positive for human immunodeficiency virus (HIV).
  18. Pregnant/lactating women, or women with the possibility of pregnancy.
  19. Individuals who have participated in other drug trials within 4 weeks.
  20. Other conditions deemed unsuitable for participation in this clinical trial by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the tolerability and safety for intravenous HNF4α srRNA in subjects with metastatic colorectal cancer | Through study completion, an average of 2 years
  Safety and tolerability are assessed based on the incidence of Dose-Limiting Toxicities (DLTs) within 14 days post-initial drug administration, along with the frequency and severity of adverse events (AEs), serious adverse events (SAEs), and events leading to treatment discontinuation throughout the treatment period, all evaluated using the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
  According to Amendment 1, the primary endpoint has been amended from assessing the incidence and severity of DLTs, adverse events (AEs), serious adverse events (SAEs), and AEs leading to treatment discontinuation (evaluated per NCI-CTCAE 5.0) with HNF4α srRNA therapy to assessing these outcomes for both HNF4α srRNA monotherapy and combination therapy.

SECONDARY OUTCOMES:
To assess the objective response rate (ORR) by RECIST v1.1 | From the first study dose date until the date of documented complete response or partial response, assessed up to 24 months.
  To assess the proportion of subjects who have best overall response of complete response or partial response at the time of data cutoff based on RECIST v1.1.
  According to Amendment 1, the secondary endpoint has also been updated from evaluating the ORR per RECIST v1.1 with HNF4α srRNA therapy to evaluating the ORR for both monotherapy and combination therapy with HNF4α srRNA per RECIST v1.1.
Duration of response based on RECIST v1.1 | up to 24 months
  To assess the time from the first documentation of complete response or partial response to the date of first documentation of disease progression or death (whichever occurs first) based on RECIST v1.1
Progression-free survival based on RECIST v1.1 | up to 24 months
  To assess the time from the first study dose date to the date of first documentation of disease progression or death(whichever occurs first) based on RECIST v1.1
Time to response based on RECIST v1.1 | up to 24 months
  To assess the time from the date of first study dose to the date of first documentation of complete response or partial response based on RECIST v1.1
Clinical benefit rate based on RECIST v1.1 | up to 24 months
  To assess the proportion of subjects who have best overall response of complete response or partial response or durable stable disease (duration of stable disease ≥ 23 weeks) based on RECIST v1.1
Overall Survival | Throughout the entire course of treatment until the end of the follow-up period, an average of 2 years
  To assess the time from the first study dose date until date of death from any cause . Subjects who are lost to follow-up and the subjects who are alive at the date of data cutoff will be censored at the date the subject was last known alive or the cut-off date, whichever comes earlier.
Patient Reported Outcome-1 | Through study completion, an average of 2 years
  the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). The maximum and minimum values of the EORTC QLQ-C30 questionnaire depend on the specific items and domains. For items with 7 levels, the maximum value is 7 points, and the minimum value is 1 point; for items with 4 levels, the maximum value is 4 points, and the minimum value is 1 point. In the standardized scores, the theoretical maximum score is 100 points, and the minimum score is 0 points. However, under normal circumstances, a higher score does not always represent a better outcome, as the interpretation of the scores needs to be based on the specific items and domains of the scale.
Patient Reported Outcome-2 | Through study completion, an average of 2 years
  Functional Assessment of Cancer Therapy Cololrectal Cancer (FACT-C). Each item has 5 levels, ranging from none to extreme. For assessments of functioning and overall health status, a higher score indeed indicates better patient conditions. However, for some symptom scales, such as pain or fatigue, a higher score actually signifies more severe issues.
Patient Reported Outcome-3 | Through study completion, an average of 2 years
  The Generic Euroquol Five Dimension Five Level (EQ-5D-5L) Questionnaire. The EQ-5D-5L includes five dimensions: Mobility, Self-care, Usual Activities, Pain/Discomfort, and Anxiety/Depression, each with 5 levels ranging from &#39;No problems&#39; to &#39;Unable to perform/Extremely severe&#39;. In addition, there is a Visual Analogue Scale (EQ VAS), which ranges from 0 (the worst health state you can imagine) to 100 (the best health state you can imagine). The EQ VAS score reflects an individual assessment of their overall health status. The scores of the EQ-5D-5L are not necessarily better when they are higher, as they reflect the individual health status relative to societal preferences.
The impact of HNF4α srRNA treatment on tumor biomarkers in serum | Through study completion, an average of 2 years
  The changes in tumor markers after treatment, including CA19-9, and carcinoembryonic antigen (CEA)

OTHER OUTCOMES:
The assessment of whether the efficacy of HNF4α srRNA is related to specific mutations | Through study completion, an average of 2 years
  Identification of whether the efficacy of HNF4α srRNA is related to specific gene mutations in CRC tissue through next-generation sequencing
The impact of HNF4α srRNA treatment on cytokines in serum | Through study completion, an average of 2 years
  The detection of cytokines in patient serum before and after treatment of HNF4α srRNA
The impact of HNF4α srRNA treatment on immune cell subsets in serum or tissuses | Through study completion, an average of 2 years
  The detection of immune cell subsets in patient serum or tissues before and after treatment of HNF4α srRNA

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Fen Xie, MD. PhD, Principal Investigator — Naval Medical University
Locations (1):
- Shanghai Changzheng Hospital，Naval Medical University, Shanghai, Shanghai Municipality, China